CLINICAL TRIAL: NCT06342037
Title: NOvel Immunotherapy Strategies for Advanced Triple Negative Breast Cancer (TNBC) Patients: TONIC-3 Trial
Acronym: TONIC-3
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N22TON
Record Dates: First submitted 2024-03-07; First posted 2024-04-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Metastatic Breast Cancer
Keywords: Triple negative breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Tiragolumab; atezolizumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Tiragolumab and atezolizumab (Experimental): Tiragolumab 600mg and atezolizumab 1200 mg, both every three weeks
  Interventions: Drug: Tiragolumab; Drug: Atezolizumab
- Tiragolumab and ipilimumab (Experimental): Tiragolumab 600mg every 3 weeks and ipilimumab 1mg/kg every 3 weeks for the first 4 cycles
  Interventions: Drug: Tiragolumab; Drug: Ipilimumab
- Tiragolumab, atezolizumab and ipilimumab (Experimental): Tiragolumab 600mg and atezolizumab 1200mg both every 3 weeks, plus ipilimumab 1mg/kg every 3 weeks for the first 4 cycles
  Interventions: Drug: Tiragolumab; Drug: Atezolizumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Tiragolumab — 600mg every 3 weeks (Q3W)
Drug: Atezolizumab — 1200mg every 3 weeks (Q3W)
  Other Names: Tecentriq
  Arms: Tiragolumab and atezolizumab; Tiragolumab, atezolizumab and ipilimumab
Drug: Ipilimumab — 1 mg/kg, maximum of 4 cycles
  Other Names: Yervoy
  Arms: Tiragolumab and ipilimumab; Tiragolumab, atezolizumab and ipilimumab

SUMMARY:
This is a single center, non-blinded, multi-cohort, non-comparative phase II trial to study the safety and efficacy of tiragolumab with atezolizumab and/or ipilimumab in advanced triple-negative breast cancer.

DETAILED DESCRIPTION:
Programmed cell death protein 1 (PD1) -blockade is currently being approved for the neoadjuvant treatment of early TNBC as well as for first-line treatment in combination with chemotherapy for patients with Programmed cell death-ligand 1 (PD-L1) -positive TNBC with metastatic disease. However, response rates are modest, responses are not always durable and PD-L1 is a suboptimal biomarker to select patients for this regimen. Therefore, the overarching goal of this TONIC-3 study is to develop novel immunomodulatory strategies for patients with advanced TNBC making use state-of-the-art research tools to better understand the underlying cancer-immune interactions of this disease

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or incurable locally advanced triple negative breast cancer with confirmation of Estrogen receptor (ER) and Human Epidermal growth factor Receptor 2 (HER2) negativity (ER <10%, HER2 IHC 0, 1+ or 2+ with no amplification) on a histological biopsy of a metastatic lesion
* Patients with PD-L1 negative disease determined using the Combined Positivity Score (CPS<10) (Dako 22C3 IHC) OR previously treated with anti-PD(L)1 in the (neo)adjuvant or metastatic setting (irrespective of PD-L1 status).
* Metastatic lesion accessible for histological biopsy
* 18 years or older
* World Health Organisation (WHO) performance status of 0 or 1
* Maximum of three lines of chemotherapy, including antibody-drug conjugates and Poly-ADP Ribose Polymerase (PARP)-inhibitors, for metastatic disease and with evidence of progression of disease
* Measurable or evaluable disease according to RECIST1.1
* Disease Free Interval (defined as time between first diagnosis or locoregional recurrence and first metastasis) longer than 1 year. This does not apply to patients with de novo metastatic disease or patients who did not receive (neo)adjuvant chemotherapy.
* Adequate bone marrow, kidney and liver function

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris
* Symptomatic brain metastases (subjects with asymptomatic brain metastases are eligible if these are free of progression for at least 4 weeks)
* History of leptomeningeal disease localization
* History of having received other anticancer therapies within 2 weeks of start of the study drug
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivy to Chinese hamster ovary cell products or to any component of the atezolizumab or tiragolumab formulation
* History of immunodeficiency, autoimmune disease, conditions requiring immunosuppression (>10 mg daily prednisone equivalents) or chronic infections.
* Prior treatment with an anti-CTLA4 or anti-TIGIT antibody.
* Administration of live vaccine within 30 days of planned start of study therapy.
* Active other cancer
* Positive test for hepatitis B, hepatitis C, HIV and/or Epstein Barr virus (EBV)
* History of uncontrolled serious medical or psychiatric illness
* Current pregnancy pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
PFS-12 | Assessed at 12 weeks
  Progression-free survival rate as measured by the proportion of patients free of progression after 12-weeks of treatment
Incidence of adverse events | Assessed until 90 days after the last dose of study treatment or until initiation of new anti-cancer therapy, whichever occurs first
  Number of patients with adverse events as measured according to CTCAE v5.0

SECONDARY OUTCOMES:
Objective response rate | Assessed at week 6, week 12 and every 12 weeks thereafter; assessed up to 120 months
  Complete response or partial response according to Response Evaluation Criteria in Solid Tumours in cancer immunotherapy trials (iRECIST) and Response Evaluation Criteria in Solid Tumours (RECIST version 1.1)
Clinical benefit rate | Assessed at week 6, week 12 and every 12 weeks thereafter; assessed up to 120 months
  Complete response, partial response or stable disease for at least 24 weeks according to iRECIST and RECIST1.1
Progression-free survival | Assessed at week 6, week 12 and every 12 weeks thereafter; median 12 months
  Time from randomization to data of first tumor progression
Overall survival | Assessed monthly until date of death; median 12 months
  Time from therapy initiation to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Marleen Kok, MD, Principal Investigator — Antoni van Leeuwenhoek
Locations (1):
- Antoni van Leeuwenhoek, Amsterdam, North Holland, Netherlands